CLINICAL TRIAL: NCT06650215
Title: Validity and Reliability of the 2-minute Walk Test in Hemodialysis Patients
Brief Title: The 2-minute Walk Test in Hemodialysis Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Kirsehir Ahi Evran Universitesi (Other)
Responsible Party: Principal Investigator, Merve Firat, Assistant Professor, Kirsehir Ahi Evran Universitesi
Other Study IDs: 2024-13/113
Record Dates: First submitted 2024-10-18; First posted 2024-10-21 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-10

CONDITIONS: End Stage Renal Disease
Keywords: Hemodialysis
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Walking tests are widely used to assess functional capacity in different populations because of their ease of administration, interpretability and representativeness of activities of daily living.The aim of our study was to investigate the validity and reliability of the 2-minute walk test in hemodialysis patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with end stage renal disease receiving hemodialysis
* Being clinically stable
* Being Aged between 18-80
* Volunteering to participate in this study

Exclusion Criteria:

* Having a musculoskeletal problem that may affect functional capacity measurement
* Having had a cardiac event in the past 3 months

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hemodialysis patients who are clinically stable, between 18 and 80 years of age, who are being followed up at the Hemodialysis Unit of Kırşehir Education and Research Hospital, who do not have any exclusion criteria, who can adapt to the evaluations to be made, who are willing to volunteer and who sign the informed consent form will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Estimated)
Dates: Start 2024-11 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Exercise capacity | 5 minutes
  Will be assessed using the 2 minute walk test.
Exercise capacity | 10 minutes
  Will be assessed using the 6 minute walk test.
Muscle functions | 1 minutes
  Will be evaluated with 1 minute sit-stand test.

SECONDARY OUTCOMES:
Physical activity | 5 minutes
  Will be evaluated using International Phsyical Activity Questionnaire-Short form

CONTACTS AND LOCATIONS:
Overall Officials: Merve Firat, Principal Investigator — Kirsehir Ahi Evran University
Locations (1):
- Kirsehir Ahi Evran University, Kırşehir, Turkey (Türkiye)